CLINICAL TRIAL: NCT04280601
Title: A Local Interventional Study in a Cohort of Patients With GPA, MPA and EGPA (PART 2 of "Vitamin D Status in ANCA-associated Vasculitis: Analysis of RDCRN-VCRC and Local Clinic Cohorts of Patients With GPA, MPA and EGPA")
Brief Title: PRagmatic Analysis of Vitamin D in ANCA-Associated Vasculitis
Acronym: PRAVDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Pagnoux (Other)
Responsible Party: Sponsor-Investigator, Christian Pagnoux, MD, MPH, MSc, Mount Sinai Hospital, Canada
Organization: Mount Sinai Hospital, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0039-E
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: ANCA-associated Vasculitis; Granulomatosis With Polyangiitis; Microscopic Polyangiitis; Eosinophilic Granulomatosis With Polyangiitis
Keywords: Vitamin D; ANCA; Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Vasculitis | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Patients with insufficient and/or deficient vitamin D status (<75 nmol/L) at study enrolment will be instructed to take a 12-month supply of vitamin D3 supplementation (to a maximum of 2,000 IU/day) vs. those with sufficient status will be observed for 12-months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low vitamin level at baseline (Other): At specific time points we will measure vitamin D status (baseline and 12-months) and re-enforcing vitamin D supplementation in those with insufficient or deficient vitamin D levels. More specifically, we will ask patients with insufficient or deficient vitamin D levels at enrollment to increase vitamin D intake by 1,000 IU units (to a maximum of 2,000 IU if the patient is already on vitamin D supplementation) for the 12 month period.
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D — Patients with insufficient and/or deficient vitamin D status (<75 nmol/L) at study enrolment will be instructed to take a 12-month supply of vitamin D3 supplementation (to a maximum of 2,000 IU/day) vs. those with sufficient status will be observed for 12-months

SUMMARY:
This prospective study will assess if 12 months of vitamin D3 (cholecalciferol) supplementation, in patients with AAV (GPA, MPA, and EGPA) who have deficient or insufficient 25(OH)D3 status at enrollment, correlates with improved disease activity and/or lower frequency of relapse (compared to historical data and a previously conducted cross sectional study (part I) that assessed vitamin D status in a cohort of similar patients).

DETAILED DESCRIPTION:
1. Subject cohorts: Patients with a diagnosis of AAV from the MSH Rheumatology clinic in a cohort of consecutive patients over a 3 month recruitment period.
2. Study Design, Data Collection: Patients with insufficient and/or deficient vitamin D status at study enrolment will be instructed to take 12 months of vitamin D3 (cholecalciferol) supplementation (1000 IU for those not on vitamin D, or to increase the dose up to 2000 IU per day for those already on vitamin D) vs. those with sufficient status who will be observed for 12-months.
3. Study Duration: 12 months.
4. Study Endpoints: Vitamin D status vs. disease activity.

ELIGIBILITY:
Inclusion criteria:

* Patients at least 18 years of age, women and men
* Followed at the Mount Sinai Hospital, Vasculitis clinic, Toronto
* With a diagnosis of AAV (GPA, MPA or EGPA) satisfying the modified American College of Rheumatology 1990 classification criteria and/or the revised 2012 Chapel Hill nomenclature definition.

Exclusion criteria:

* Current or history of hypercalcemia, primary hyperparathyroidism, sarcoidosis, hypervitaminosis D, Williams syndrome, other autoimmune, chronic inflammatory or infectious conditions, malabsorptive disorders, cancer, type 1 diabetes, liver disease
* Current or planned pregnancy within the next year.
* Intolerance, allergy to oral vitamin D, and/or contra-indication to take oral vitamin D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Disease activity and disease relapse (using BVAS) | 12 months
  Number of patients with active disease (BVAS score) or disease relapse (new item on the BVAS, in patients previously in remission) between enrollment and month 12, according to the study arm intervention (normal baseline vitamin D level vs. low baseline level and asked to increase vitamin D intake)

SECONDARY OUTCOMES:
Renal function (GFR) | 12 Months
  Number of patients with progressive renal AAV-related disease (worsening GFR) in each study arm between enrollments and month 12
Cardiovascular events | 12 Months
  Number of patients with cardiovascular events (IM, stroke) in each study arm between enrollments and month 12
Interstitial lung disease diagnosis or progression (imaging and PFT) | 12 Months
  Number of patients with new diagnosis of ILD or worsening of ILD in each study arm (based on clinical, and either imaging and/or PFT findings) between enrollments and month 12
Glucocorticoid use (and cumulative dose, mg) | 12 months
  Use of glucocorticoids (including cumulative dose) in each study arm between enrollment and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pagnoux, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Vasculitis clinic, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the Canadian vasculitis research network, listing ongoing studies and their status in Canada — http://www.canvasc.ca